CLINICAL TRIAL: NCT04493528
Title: Needle-free Dental Anesthesia: a Pilot Split-mouth Cross-over Randomized Clinical Trial.
Brief Title: Needle-free Dental Anesthesia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: MEDICAL INTERNATIONAL TECHNOLOGIES (MIT CANADA) INC. (Unknown)
Responsible Party: Principal Investigator, Faleh Tamimi, Associate Professor, Accociate Dean, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A09-M36-18A
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia, Local; Needle Phobia
Keywords: Needle-free injection; Dental anesthesia; Infiltration; Nerve block

STUDY DESIGN:
Intervention Model Description: Randomized split-mouth cross-over clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Each participant receive two anesthesia methods randomly. Total 8 arms, 4 groups, each group will recruit 6 participants. Incase of drop out, a total of 30 participant will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Needle Infiltration anesthesia (Active Comparator): Patients received one needle injection of infiltration anesthesia at left or right upper lateral incisors using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Needle,2% lidocaine(xylocaine)
- Needle-free infiltration anesthesia (Experimental): Patients received one NFLJI (needle-free liquid jet injection) of infiltration anesthesia at left or right upper lateral incisors using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Meso-Jet, 2% lidocaine(xylocaine)
- Needle mental nerve block (Active Comparator): Patients received one needle injection of mental nerve block at left or right lower premolar region using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Needle,2% lidocaine(xylocaine)
- Needle-free mental nerve block (Experimental): Patients received one NFLJI (needle-free liquid jet injection) of mental nerve block at left or right lower premolar region using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Meso-Jet, 2% lidocaine(xylocaine)
- Needle mandibular nerve block (Active Comparator): Patients received one needle injection of mandibular nerve block at left or right mandibular foramen using 2 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Needle,2% lidocaine(xylocaine)
- Needle-free mandibular nerve block (Experimental): Patients received one NFLJI (needle-free liquid jet injection) of mandibular nerve block at left or right mandibular foramen using 2 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Meso-Jet, 2% lidocaine(xylocaine)
- Needle infraorbital nerve block (Active Comparator): Patients received one needle injection of infraorbital nerve block at left or right canine fossa using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Needle,2% lidocaine(xylocaine)
- Needle-free infraorbital nerve block (Experimental): Patients received one NFLJI (needle-free liquid jet injection) of infraorbital nerve block at left or right canine fossa using 1 ml 2% lidocaine with 1:50,000 epinephrine (xylocaine).
  Interventions: Combination Product: Meso-Jet, 2% lidocaine(xylocaine)

INTERVENTIONS:
Combination Product: Meso-Jet, 2% lidocaine(xylocaine) — Performing local dental anesthesia using needle-free liquid jet injection with different parameters (pressure, volume, injection technique). Anesthetic agent: 2% lidocaine with 1:100,000 epinephrine, dose: 0.3-2ml.
  Other Names: needle-free device; jet injector; NFLJI (Needle-free liquid jet injection system)
  Arms: Needle-free infiltration anesthesia; Needle-free infraorbital nerve block; Needle-free mandibular nerve block; Needle-free mental nerve block
Combination Product: Needle,2% lidocaine(xylocaine) — Performing local dental anesthesia using syringe and needles, same as regular clinical practice. Anesthestic agent: 2% lidocaine with 1:100,000 epinephrine,dose: 0.3-2ml.
  Arms: Needle Infiltration anesthesia; Needle infraorbital nerve block; Needle mandibular nerve block; Needle mental nerve block

SUMMARY:
Many patients experience pain and anxiety from traditional needle anesthesia and may avoid necessary dental treatments. The needle-free liquid jet injection(NFLJI) could solve these problems. NFLJI delivers drug solutions by creating a micro-thin pressure liquid jet to penetrate the skin and disperse in the soft tissue. It has many advantages like eliminating injection pain, needle phobia and needle disposal. However, anesthesia techniques in dentistry were all developed for needle injection, and they are not very effective for NFLJI. Moreover, clinical trials of dental anesthesia using NFLJI have shown inconsistent efficacy.

In this study, we aim to compare the clinical efficacy between NFLJI and needle dental anesthesia in pilot split-mouth cross-over randomized clinical trials, assess the feasibility to conduct such trial on a larger scale.

Participants will be assigned to one of the following four groups: 1. Infiltration on a maxillary lateral incisor,2. Inferior alveolar nerve block, 3.Mental nerve block, 4. Infraorbital nerve block. Each participant will receive one injection with a needle and another one with NFLJI randomly at the same appointment. A washout period of 1 hour between two procedures for participants' to forget the previous experience. Needle injection will be performed according to clinical standards. NFLJI will be performed according to a guideline developed in our research group. Participants will stay in the clinic until the anesthesia effect disappear and be followed for one week.

The primary outcome is the efficacy and effect of two anesthesia interventions. The secondary outcome is the pain and anxiety visual analogue scale before and during injection, taste preference, and complications. Additionally, patients' overall feelings for two interventions as well as any barriers to conducting such a trial will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-35 years-old
* fluent in English
* cooperate

Exclusion Criteria:

* has a history of chronic pain,
* has a systematic disease,
* has root canal therapy at the upper lateral incisor/lower posterior teeth region.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Dental pulp anesthesia | 10 minutes after injection.
  Dental pulp anesthesia result is measured by an electric pulp test(EPT), successful anesthesia for dental pulp exhibits an EPT at 80.
Efficacy of dental pulp anesthesia | 10 minutes after injection.
  The number of sucessful dental pulp anesthesia cases over total number of participants in the group.
Time to initiation of anesthesia | 1 minute after injection
  Time to initiation of anesthesia feeling, measured by a simple pinch test using a periodontal probe
Time to termination of anesthesia | 3 hours after injection
  Time to termination of anesthesia feeling, measured by a simple pinch test using a periodontal probe

SECONDARY OUTCOMES:
Baseline pain level | 1 minute before injection
  Participants' pain level before receiving the needle or needle-free injection, measured by standard visual analog scale for pain. From 0 to 10, 0 stands for "no pain", 10 stands for "worst pain". Higher score means a worse outcome.
Pain level during injection | 10 seconds after the injection
  Participants' pain level when receiving the needle or needle-free injection, measured by standard visual analog scale for pain. From 0 to 10, 0 stands for "no pain", 10 stands for "worst pain". Higher score means a worse outcome.
Baseline anxiety level | 1 minute before injection
  Participants' anxiety level before receiving the needle or needle-free injection, measured by visual analogue scale for anxiety. From 0 to 10, 0 stands for ""Not at all Anxious", 10 stands for "Extremely Anxious". Higher score means a worse outcome.
Anxiety level during injection | 10 seconds after the injection.
  Participants' anxiety level when receiving the needle or needle-free injection, measured by visual analogue scale for anxiety.From 0 to 10, 0 stands for ""Not at all Anxious", 10 stands for "Extremely Anxious". Higher score means a worse outcome.
Taste preference | 1 minute after the injection
  Participants' taste preference after needle or needle-free injection, measured by 9-point hedonic scale for measuring food acceptability. From 1 to 9, 1 stands for "dislike extremely", 5 stands for "neither like or dislike", 9 stands for "like extremely". Higher score means a better outcome.
Incidence of adverse effect [safety] | 10 seconds after injection.
  Incidence of adverse effect immediately after aneshesia injection, such as tissue damage, bleeding, hematoma.
Incidence of adverse effect during follow-up period[safety] | up to 7 days
  Incidence of adverse effect after aneshesia procedure during follow-up period, such as: ulcer, hematoma, discomfort, abnormal feeling, nerve damage.

OTHER OUTCOMES:
Participant's feedbacks | 20 minutes after all procedures.
  Reord participants's feedbacks about the whole trial, such as: overall feelings, preferences,complains.
Barriers | through study completion, from date of recruitment until the date of last follow-up case complition, an average of 6 month.
  Record possible barriesrs in recruitment,randomization,operation.

CONTACTS AND LOCATIONS:
Overall Officials: Faleh Tamimi, Ph.D., Principal Investigator — McGill University Faculty of Dentistry
Locations (1):
- McGill University Faculty of Dentistry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No